CLINICAL TRIAL: NCT05645237
Title: Health-Related Quality of Life in Prostate Cancer Patients Treated With Radiotherapy
Brief Title: HRQOL in Prostate Cancer Patients Treated With Radiotherapy
Acronym: PRORAD
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Wilma Heemsbergen, Clinical Epidemiologist, Project Leader, PhD, Erasmus Medical Center
Other Study IDs: MEC-2018-1711; project nr 14259 (HYPROSTAR) (Other Grant/Funding Number: Dutch Cancer Society (KWF))
Record Dates: First submitted 2022-11-28; First posted 2022-12-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radiotherapy; hypofractionation; health-related quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Applied radiotherapy protocol (subcohort) 1: 60 Gy in 20 fractions of 3 Gy external beam radiotherapy
  Interventions: Radiation: radiotherapy
- Applied radiotherapy protocol (subcohort) 2: 42.7 Gy in 7 fractions of 6.1 Gy external beam radiotherapy
  Interventions: Radiation: radiotherapy
- Applied radiotherapy protocol (subcohort) 3: 38 Gy in 4 fractions of 9 Gy stereotactic external beam radiotherapy
  Interventions: Radiation: radiotherapy
- Applied radiotherapy protocol (subcohort) 4: 27 Gy in 2 fractions of 13.5 Gy brachytherapy
  Interventions: Radiation: radiotherapy
- Applied radiotherapy protocol (subcohort) 5: 72 Gy in 36 fractions of 2 Gy postoperative external beam radiotherapy
  Interventions: Radiation: radiotherapy
- Applied radiotherapy protocol (subcohort) 6: 70 Gy in 35 fractions of 2 Gy on prostate combined with 52 Gy in 28 fractions of 2 Gy on pelvic lymph node areas, external beam radiotherapy.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy is delivered with linear accelerators or cyberknife (external beam radiotherapy), or local irradiation with high dose rate brachytherapy (brachytherapy)

SUMMARY:
The study primarily aims at evaluating health-related quality of life after radiotherapy for prostate cancer, using modern hypofractionated radiotherapy schedules. Study design is a prospective observational cohort study. All patients give written informed consent and fill out online validated questionnaires before, during, and after radiotherapy (yearly) up to 5 years post-treatment.

DETAILED DESCRIPTION:
Rationale: Patient-Reported Outcomes (PROs), such as health-related quality of life (HRQL), have achieved an important role in the evaluation of benefits and harms after cancer treatment, including radiotherapy for prostate cancer (PCa). In the past year, clinical radiotherapy protocols at the Erasmus MC have been changed for external beam radiotherapy (EBRT) as well as for brachytherapy (BT). In order to evaluate the current, changed, clinical practice, we will conduct a prospective cohort study, with the main purpose to assess HRQL for the current treatment options at the Erasmus MC.

Objective: To establish HRQL (start treatment - 5 years after treatment) in a prospective cohort of ≈600 patients with localized PCa treated with radiotherapy within in the period ≈ 1/3/2019 - 1/12/2023.

Main objective: to establish changes in HRQL levels (with respect to baseline) up to 5 year post-treatment, within each radiotherapy modality for prostate cancer patients, i.e. EBRT 60 Gy in 20 fractions, EBRT 42.7 Gy in 7 fractions, CyberKnife (stereotactic EBRT) 38 Gy in 4 fractions, BT 27 Gy in 2 fractions, postoperative EBRT (PORT) 72 Gy in 36 fractions, EBRT for LN+: 70 Gy (prostate)/52 Gy (lymph nodes) in 28 fractions.

Study design: Prospective observational cohort study. Study population: Patients with prostate cancer T1c-T4 referred for radiotherapy at the Erasmus MC as a primary treatment with curative intent or as first line adjuvant treatment after a prostatectomy.

Intervention: All interventions are according to applicable standard clinical procedures & protocols for localized prostate cancer of the Radiotherapy department.

Main study parameters/endpoints: HRQL scores of the EPIC (urinary domain, bowel domain), and the IIEF-5 (sexual function) score.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no additional risks or benefits for patients that participate in the study. The additional burden is to fill out questionnaires at regular intervals.

Study patient recruitment period was from April 2019 to May 2025, enrolling about 695 eligible patients, mainly treated with UHF 7x6.1 Gy (n=240), MHF 20x3/3.1 Gy (n=210), PORT (n=85), and brachytherapy (n=65).

ELIGIBILITY:
Inclusion Criteria:

* Clinically T1c-T4, N0 (or N+ in case of EBRT-LN+), M0 prostate cancer patient referred for radiotherapy.
* Willing and capable to fill out Dutch questionnaires on health-related items at a computer (online questionnaires).
* Signed written Informed Consent.

Exclusion Criteria:

* Previously radiation treatment in the pelvic region, for any reason.
* Diagnosed with other tumor in the past 12 months or known with tumor progression of another tumor.
* Postoperative radiotherapy with dose levels < 72 Gy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinically T1c-T4, N0 (or N+ in case of EBRT-LN+), M0 prostate cancer patients referred for radiotherapy to the Erasmus Medical Center.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
EPIC questionnaire score on urinary domain | Year 1 - Year 4
  Expanded Prostate Cancer Index Composite (EPIC) Urinary Domain score: a 0 to 100 scale with higher scores representing better HRQOL.
EPIC questionnaire score on bowel domain | Year 1 - Year 4
  Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain score: a 0 to 100 scale with higher scores representing better HRQOL.
Sexual functioning score on IIEF-5 questionnaire | Year 1- Year 4
  Sexual functioning score on International Index of Erectile Function (IIEF-5) questionnaire: 1 to 25 scale, higher scores imply better function

SECONDARY OUTCOMES:
Acute rectal bleeding, on symptom checklist (patient-reported) | During radiotherapy - 3 months after radiotherapy
  Rectal bleeding is scored on a symptom checklist on a Likert scale (bother: none, little, quite, a lot) (patient-reported), higher score means worse symptoms. This symptom checklist was locally developed and used in previous trials.
Acute mucous discharge, on symptom checklist (patient-reported) | During radiotherapy - 3 months after radiotherapy
  Mucous discharge is scored on a symptom checklist on a Likert scale (bother: none, little, quite, a lot) (patient-reported), higher score means worse symptoms. This symptom checklist was locally developed and used in previous trials.
Late moderate to severe urinary incontinence | Year 1 - Year 4
  Score of 'more than once a week or daily leaking of urine' on the Expanded Prostate Cancer Index Composite (EPIC) Urinary Domain.
Late moderate to severe urinary frequency during the night | Year 1 - Year 4
  Score of 'moderate/big problem for waking up to urinate' on the Expanded Prostate Cancer Index Composite (EPIC) Urinary Domain.
Late moderate to severe incontinence for stools | Year 1 - Year 4
  Score of 'more than once a week or daily uncontrolled leakage of stools/feces' on the Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain.
Late frequent bowel movements | Year 1 - Year 4
  Score of 'more than five' daily bowel movements on the Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain.
Late erectile dysfunction | Year 1- Year 4
  Score of 'very low/low confidence to get and keep an erection' on the International Index of Erectile Function (IIEF-5) questionnaire.

OTHER OUTCOMES:
General health score on EQ-5D-5L questionnaire | Year 1- Year 4
  General health score on EuroQoL 5-dimensions, 5-levels (EQ-5D-5L) questionnaire: total score between -1 - +1,higher score indicates better quality of life.
Acute moderate to severe rectal discomfort | During radiotherapy - 3 months after radiotherapy
  Score of 'quite/a lot' for the symptom 'pain with stools' and/or 'cramping urge',
Late watery bowel movements | Year 1 - Year 4
  Score of 'moderate/big problem for watery bowel movements' on the Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain.
Late gastrointestinal pain | Year 1 - Year 4
  Score of 'moderate/big problem for abdominal/pelvic/rectal pain' on the Expanded Prostate Cancer Index Composite (EPIC) Bowel Domain.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Incrocci, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Radiotherapy, Erasmus MC Cancer Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Datasets used for publications (in the future) will be made available upon request. Requests for taking part in meta-analyses initiated by other research groups will be considered after publication of the main endpoints.

REFERENCES:
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Utomo E, Blok BF, Pastoor H, Bangma CH, Korfage IJ. The measurement properties of the five-item International Index of Erectile Function (IIEF-5): a Dutch validation study. Andrology. 2015 Nov;3(6):1154-9. doi: 10.1111/andr.12112. Epub 2015 Oct 9. PMID 26453539
- See also: Protocol Registration Quality Control Review Criteria of ClinicalTrials.gov — https://prsinfo.clinicaltrials.gov/ProtocolDetailedReviewItems.pdf